CLINICAL TRIAL: NCT05774847
Title: Behavioral Evidence on the Modulators of Unconscious Processing in Decision-making
Brief Title: Unconscious Processing in Decision-making
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Istituto Universitario di Studi Superiori Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 2138
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: decision-making; unconscious processing; subliminal processing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All healthy participants: Healthy participants will be recruited and assigned to different behavioral studies assessing the effect of the experimental manipulations of interest on decision-making metrics.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This behavioral study on healthy participants aims to provide a baseline reference for assessing alterations of decision-making performance in pathological conditions. To this purpose, this single center non-interventional behavioral study will assess the extent to which decision-making performance is affected by distinct experimental manipulations, as well as by ageing effects, in 200 healthy individuals. The main questions it aims to answer are:

* to what extent is decision-making performance stable, within individuals, regardless of non-economic manipulations concerning stimuli perceptual features as well as type of processing and motor response required to participants?
* are these manipulations additionally influenced by participants' age?

Healthy participants will be recruited for distinct behavioral studies assessing the effects of the aforementioned manipulations of distinct metrics of decision-making performance, such as loss aversion, risk aversion, and delay discounting.

DETAILED DESCRIPTION:
The fast growth of so-called Decision Neuroscience has clearly shown the implications of methods and results from behavioral economics as a potential bridge for translational research in neuro-psychiatric settings. The combination of behavioral and neural metrics allows to describe decision-making across multiple levels of explanation ranging from biological dispositions to contextual influences. To date, however, the translational implications of Decision Neuroscience are constrained by a relatively limited knowledge of the potential modulators of decision-making, which seem to include perceptual, cognitive and motor variables. In this regard, there is largely sparse evidence concerning the modulation of choices by highly different factors such as a) perceptual features of the stimuli (e.g., spatial distance between visually-presented potential gains and losses); b) type of processing required to participants (e.g., select vs. reject an option); c) type of motor response required to communicate the decision (e.g., press vs. release a button); d) subliminal vs. supraliminal perception of the stimuli. Moreover, there is evidence of ageing effects on decision-making, particularly when choice-related evaluations involve a trade-off between reward and risk. On this ground, this single center non-interventional behavioral study aims to investigate whether, and how, distinct well-established metrics of decision-making are influenced by the aforementioned factors. To this purpose, 200 healthy individuals will be recruited and assigned to different behavioral studies aimed to assess the effect of the aforementioned manipulations on well-established gambling tasks resulting in individual metrics of loss aversion (the tendency to prefer avoiding losses to acquiring equivalent gains), risk aversion (the preference for certain outcomes over probabilistic ones), and delay discounting (the decline in the present value of a reward with delay to its receipt). The results of this study are expected to provide a baseline reference for assessing alterations of decision-making performance in pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, as determined by screening assessments and principal investigator judgment
* The participant must be able to comply with study requirements as judged by the principal investigator

Exclusion Criteria:

* Any history of alcohol and/or drug abuse, addiction or suspicion of regular consumption of drugs of abuse
* Use of any psychoactive medication, or medications known to have effect on central nervous system

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 200 healty individuals, aged 18-60 years, sampled from the general population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Individual index of loss aversion | Behavioral-study day 1
  This variable reflect the spontaneous disposition to overweigh potential losses, compared with equivalent gains in decision-making, resulting in the tendency to avoid potential losses more than approach potential gains.

SECONDARY OUTCOMES:
Individual index of risk aversion | Behavioral-study day 1
  This variable reflect the spontaneous preference for certain, compared with probabilistic, outcomes, resulting in the tendency to avoid risky options regardless of their expected value.
Individual index of delay discounting | Behavioral-study day 1
  This variable reflects the tendency to discount delayed utilities/rewards compared with immediate ones, resulting in choices driven by the impulsive search for immediate gains regardless of potential larger future outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Ita, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Requests for sharing will assessed case by case, and data will be made available on reasonable request.